CLINICAL TRIAL: NCT00831064
Title: A Randomized Controlled Trial of Four Different Bowel Cleansing Regimens Prior to Colonoscopy: Efficacy, Patient Tolerability and Safety
Brief Title: A Trial of Four Different Bowel Cleansing Regimens Prior to Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Dina Kao, Associate Professor, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 1-Kao
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-06

CONDITIONS: Bowel Preparation
Keywords: bowel preparation quality; colonoscopy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1. 4L PEG only (Active Comparator): 4L PEG PO
  Interventions: Procedure: colonoscopy bowel prep
- 2. 2L PEG plus bisacodyl (Active Comparator): 2L PEG PO + 4 tablets bisacodyl PO
  Interventions: Procedure: colonoscopy bowel prep
- 3. NaP (Active Comparator): 90 cc NaP PO
  Interventions: Procedure: colonoscopy bowel prep
- 4. PSMC plus Mg-citrate (Active Comparator): PSMC plus 300 cc Mg-citrate PO
  Interventions: Procedure: colonoscopy bowel prep

INTERVENTIONS:
Procedure: colonoscopy bowel prep — PEG, bisacodyl, NaP, PSMC and Mg-citrate

SUMMARY:
To compare 4 commonly used bowel preparations in terms of efficacy, patient tolerability and safety. All these 4 bowel preparations are likely to be efficacious and safe. However, those with lower volume are likely to be better tolerated and completed by patients.

DETAILED DESCRIPTION:
Adequate bowel preparation is imperative for diagnostic accuracy and therapeutic safety. Several bowel cleansing preparations have been approved by Health Canada and are commonly used prior to colonoscopy. Polyethylene glycol (PEG) has been considered to be the "gold standard" for bowel preparation. It is a nonabsorbable solution which passes through the bowel without net absorption or secretion. Significant fluid and electrolyte shifts are therefore avoided. However, the large volume (4 liters), the salty taste and the sulphur smell frequently lead to poor tolerability and compliance, sometimes resulting in inadequate bowel preparation. Several other bowel cleansing preparations have been developed and include sodium phosphate (NaP), magnesium citrate, and sodium picosulphate plus magnesium oxide (PSMC)-containing preparations. NaP is a low volume hyperosmotic solution which draws plasma water into the bowel lumen to promote colonic cleansing. As a result, significant fluid and electrolyte shifts can occur. The advantage of the low volume is better patient tolerance compared to PEG. However, even in healthy individuals severe electrolyte disturbances have been reported when the 2 required doses are taken 12 hours apart. Therefore Health Canada has recommended that 2 doses of NaP be taken 24 hours apart. Patients with renal failure, congestive heart failure and liver failure should avoid this preparation (Grade I A). PSMC is a hyperosmotic saline laxative which increases intraluminal volume resulting in increased intestinal motility. Magnesium, a constituent of PSMC, stimulates the release of cholecystokinin which also stimulates intestinal motility. Since magnesium is eliminated by the kidney, patients with renal insufficiency or failure should also avoid this preparation.

Many randomized controlled trials have compared the efficacy and tolerability of various bowel cleansing regimens. Studies comparing full-volume (4 liters) PEG with low-volume (2 liters) PEG combined with magnesium citrate or bisacodyl have demonstrated equal efficacy of colonic cleansing but with improved patient tolerance. However, there is little data on how low volume PEG compares with NaP. The only meta-analysis of twenty nine trials on optimal bowel preparation concluded that NaP was more effective in bowel cleansing than 4-liter PEG or PSMC. However, there were only three trials comparing NaP to PSMC that met inclusion and exclusion criteria in this meta-analysis and the results have been conflicting. Also there were only three trials comparing PEG to PSMC in this meta-analysis with inconclusive data. Moreover, the mean number of patients per trial was small at 223, with the highest number of patients in a trial at 500.

A consensus document prepared by three leading American gastrointestinal societies (American Society of Gastrointestinal Endoscopy, American Society of Colon and Rectal Surgeons and Society of American Gastrointestinal and Endoscopic Surgeons) as well as a position paper by the Canadian Association of Gastroenterology identified the lack of an ideal bowel preparation which meets all these criteria. Furthermore, the need for further studies was identified in the following areas:

1. Two-liter PEG vs NaP
2. PSMC vs NaP

Outpatients who need to undergo routine colonoscopy will be recruited. Each patient will be randomly assigned to one of the four bowel preparations after they have given consent to participate in the study:

1. Group 1. 4L PEG.
2. Group 2. 2L PEG plus 4 tablets of bisacodyl.
3. Group 3. 90 cc NaP.
4. Group 4. PSMC plus 1 bottle of Mg-citrate (300 cc).

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 18 and 75.
* Planned elective outpatient colonoscopy.

Exclusion Criteria:

* History of renal insufficiency or abnormal creatinine clearance with GFR <59.
* History of congestive heart failure.
* History of acute coronary syndrome or unstable angina.
* History of liver cirrhosis or ascites.
* Chronic lasix therapy.
* History of colorectal resection.
* Known or suspected bowel obstruction, megacolon or ileus

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-09; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
bowel preparation quality as measured by the Ottawa scale | at the time of endoscopy

SECONDARY OUTCOMES:
electrolyte and renal function abnormalities | 2 sets of measurements will be obtained: prior to the start of bowel preparation and at the time of colonoscopy
patient tolerability of bowel preparation | at the time of colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Sander van Zanten, MD, Study Director — University of Alberta; Din a Kao, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Sharma VK, Chockalingham SK, Ugheoke EA, Kapur A, Ling PH, Vasudeva R, Howden CW. Prospective, randomized, controlled comparison of the use of polyethylene glycol electrolyte lavage solution in four-liter versus two-liter volumes and pretreatment with either magnesium citrate or bisacodyl for colonoscopy preparation. Gastrointest Endosc. 1998 Feb;47(2):167-71. doi: 10.1016/s0016-5107(98)70351-7. PMID 9512283
- [Background] Rostom A, Jolicoeur E. Validation of a new scale for the assessment of bowel preparation quality. Gastrointest Endosc. 2004 Apr;59(4):482-6. doi: 10.1016/s0016-5107(03)02875-x. PMID 15044882
- [Background] American Society of Colon and Rectal Surgeons (ASCRS); American Society for Gastrointestinal Endoscopy (ASGE); Society of American Gastrointestinal and Endoscopic Surgeons (SAGES); Wexner SD, Beck DE, Baron TH, Fanelli RD, Hyman N, Shen B, Wasco KE. A consensus document on bowel preparation before colonoscopy: prepared by a Task Force from the American Society of Colon and Rectal Surgeons (ASCRS), the American Society for Gastrointestinal Endoscopy (ASGE), and the Society of American Gastrointestinal and Endoscopic Surgeons (SAGES). Surg Endosc. 2006 Jul;20(7):1161. doi: 10.1007/s00464-006-3037-1. No abstract available. PMID 16799744
- [Background] Rostom A, Jolicoeur E, Dube C, Gregoire S, Patel D, Saloojee N, Lowe C. A randomized prospective trial comparing different regimens of oral sodium phosphate and polyethylene glycol-based lavage solution in the preparation of patients for colonoscopy. Gastrointest Endosc. 2006 Oct;64(4):544-52. doi: 10.1016/j.gie.2005.09.030. PMID 16996347
- [Background] Schmidt LM, Williams P, King D, Perera D. Picoprep-3 is a superior colonoscopy preparation to Fleet: a randomized, controlled trial comparing the two bowel preparations. Dis Colon Rectum. 2004 Feb;47(2):238-42. doi: 10.1007/s10350-003-0027-4. PMID 15043296
- [Background] Barkun A, Chiba N, Enns R, Marcon M, Natsheh S, Pham C, Sadowski D, Vanner S. Commonly used preparations for colonoscopy: efficacy, tolerability, and safety--a Canadian Association of Gastroenterology position paper. Can J Gastroenterol. 2006 Nov;20(11):699-710. doi: 10.1155/2006/915368. PMID 17111052
- [Background] Hookey LC, Vanner S. A review of current issues underlying colon cleansing before colonoscopy. Can J Gastroenterol. 2007 Feb;21(2):105-11. doi: 10.1155/2007/634125. PMID 17299615
- [Background] Poon CM, Lee DW, Mak SK, Ko CW, Chan KC, Chan KW, Sin KS, Chan AC. Two liters of polyethylene glycol-electrolyte lavage solution versus sodium phosphate as bowel cleansing regimen for colonoscopy: a prospective randomized controlled trial. Endoscopy. 2002 Jul;34(7):560-3. doi: 10.1055/s-2002-33207. PMID 12170410
- [Background] Frommer D. Cleansing ability and tolerance of three bowel preparations for colonoscopy. Dis Colon Rectum. 1997 Jan;40(1):100-4. doi: 10.1007/BF02055690. PMID 9102248